CLINICAL TRIAL: NCT06414005
Title: A Multi-center, Randomized, Double Blinded, Placebo-controlled, Phase 2b/3 Clinical Trial to Evaluate the Safety and Efficacy of TPX-115 in Patients With Partial-thickness Rotator Cuff Tear
Brief Title: A Phase 2b/3 Study of TPX-115 on Partial-thickness Rotator Cuff Tear
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-TPX-115-22-02
Record Dates: First submitted 2024-05-10; First posted 2024-05-14 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-03

CONDITIONS: Partial Thickness Rotator Cuff Tear
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPX-115 (Experimental): Subjects receive ultrasound-guided intratendinous injection of TPX-115
  Interventions: Biological: TPX-115
- Placebo (Saline) (Placebo Comparator): Subjects receive ultrasound-guided intratendinous placebo injection
  Interventions: Other: Placebo (Saline)

INTERVENTIONS:
Biological: TPX-115 — Ultrasound-guided intratendinous injection of allogeneic fibroblasts (TPX-115)
  Arms: TPX-115
Other: Placebo (Saline) — Ultrasound-guided intratendinous placebo injection
  Arms: Placebo (Saline)

SUMMARY:
Rotator cuff tear is one of the most common shoulder diseases and conservative treatment is commonly used for tears involving ≤50% of tendon thickness. Since conventional conservative treatments are not fundamental to repair tendon tissue, there is a growing need of new therapy to improve structural outcome. This study assesses the safety and efficacy of allogeneic fibroblasts on partial-thickness rotator cuff tear. The primary outcome is change in Constant Score (CS) at 24 weeks after TPX-115 injection. Secondary outcomes include changes from baseline in CS, Visual Analogue Score (VAS) pain score, American Shoulder and Elbow Surgeons (ASES) score, Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH), Simple Shoulder Test (SST), and functional evaluations including Range of Motion (ROM) at 4, 12, 24 and 52 weeks after administration and structural evaluation using MRI at 24 and 52 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Be 19 years of age or older.
2. Have partial-thickness rotator cuff tear, ≤50% of tendon thickness or of Ellman grade II assessed by MRI.
3. Have unilateral shoulder pain, muscle weakness and limited active range of motion lasting more than 3 months despite conservative treatment
4. VAS pain score ≥4 at screening.
5. Understand fully the study and voluntarily sign the informed consent for participation in the study.

Exclusion Criteria:

1. Regardless of partial-thickness rotator cuff tear, have full-thickness rotator cuff tear confirmed by MRI.
2. Have been treated with the following

   * Have had painkiller within 1 week prior to screening visit.
   * Have had received systemic steroid or immunosuppressive agents within 4 weeks prior to screening visit.
   * Have had subacromial or intra-articular injections on the affected shoulder within 3 months prior to screening visit.
   * Have shoulder surgery on the rotator cuff tear or had received drug that included growth factor, within 6 months prior to screening visit.
3. Have been diagnosed with the following diseases.

   * Inflammatory joint diseases
   * Other shoulder diseases which may cause shoulder pain or functional disorder
   * Autoimmune diseases
   * Active hepatitis B or C
   * HIV Ab positive
   * Malignant tumors within the last 5 years
   * Coagulopathy
   * Genetic disorders related to fibroblasts of collagen
   * Other serious diseases deemed to affect the results of the study
4. Have allergies to bovine proteins or gentamicin.
5. Be pregnant, breastfeeding, planning pregnancy or unwilling to use of contraceptive suggested in this study.
6. Have participated in other clinical trials and received investigational agents within 4 weeks of this study.
7. Be deemed inadequate for the study by investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in shoulder score of Constant score (CS) | 24 weeks
  The CS total score (100) = Pain (15) + Activity of Daily Living (20) + Mobility (40) + Strength(25)

SECONDARY OUTCOMES:
Change in shoulder score of Constant score (CS) | 4, 12, 52 weeks
  The CS total score (100) = Pain (15) + Activity of Daily Living (20) + Mobility (40) + Strength(25).
hange in pain score of Visual Analogue Scale (VAS) | 4, 12, 24, 52 weeks
  VAS pain score is measured on a scale of 0 (no pain) to 10 (worst pain imaginable).
Change of American Shoulder and Elbow Surgeons (ASES) Shoulder Score | 4, 12, 24, 52 weeks
  ASES shoulder score is derived from the visual analogue scale score for pain and the activities of daily living score. The total score(100 maximum points) is weighted 50% for pain and 50% for function.
Change of Quick Disabilities of the Arm, Shoulder and Hand (Quick-DASH) Outcome Measure | 4, 12, 24, 52 weeks
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
Change in Simple Shoulder Test (SST) Score | 4, 12, 24, 52 weeks
  SST assesses functional disability of the shoulder (function related to pain, function/strength and Range of Motion).
Change in Range of Motion (ROM) | 4, 12, 24, 52 weeks
  Measurement of ROM for forward elevation, external rotation at 90º abduction, external rotation at side and internal rotation at back.
Change in Ellman grade on Magnetic Resonance Image (MRI) | 24, 52 weeks
  Ellman grade is assessed by an independent evaluator.
Change of tendinosis on MRI | 24, 52 weeks
  Tendinosis is assessed with tendinosis grading system by an independent evaluator. (0: normal, 1: mild, 2: moderate, 3: marked)

CONTACTS AND LOCATIONS:
Overall Officials: Joo Han Oh, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul